CLINICAL TRIAL: NCT01241591
Title: A Phase 3, Multi Site, Randomized, Double Blind, Placebo Controlled, Parallel Group Study Of The Efficacy And Safety Of 2 Oral Doses Of CP- 690,550 And 1 Subcutaneous Dose Of Etanercept In Subjects With Moderate To Severe Chronic Plaque Psoriasis
Brief Title: A Phase 3, Multi Site, Randomized, Double Blind, Placebo Controlled Study Of The Efficacy And Safety Comparing CP- 690,550 And Etanercept In Subjects With Moderate To Severe Chronic Plaque Psoriasis
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: A3921080
Record Dates: First submitted 2010-11-12; First posted 2010-11-16 (Estimated); Results first posted 2014-05-07 (Estimated); Last update posted 2018-12-26 (Actual); Status verified 2018-12

CONDITIONS: Psoriasis
Keywords: CP-690,550; Etanercept; Moderate; Severe; Chronic; Plaque; Psoriasis; Efficacy; Safety; Tofacitinib; Xeljanz; OPT Compare; OPT; head-to-head; non-inferiority; Psoriasis vulgaris; short-term; Itch; Pruritus; Plaque psoriasis; DLQI
MeSH Terms: conditions — Psoriasis; Lymphoma, Follicular; Bronchiolitis Obliterans Syndrome; Plaque, Amyloid; Pruritus | interventions — tofacitinib; Etanercept

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- CP 690,550 5 mg BID+Placebo BIW (Experimental)
  Interventions: Drug: CP 690,550 5 mg
- CP 690,550 10 mg BID+Placebo BIW (Experimental)
  Interventions: Drug: CP 690,550 10 mg
- Placebo BID+Etanercept 50 mg BIW (Active Comparator)
  Interventions: Biological: Etanercept 50 mg
- Placebo BID+Placebo BIW (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: CP 690,550 5 mg — CP-690,550 5 mg orally dosed twice daily and placebo subcutaneously dosed twice weekly for 12 weeks
  Arms: CP 690,550 5 mg BID+Placebo BIW
Drug: CP 690,550 10 mg — CP-690,550 10 mg orally dosed twice daily and placebo subcutaneously dosed twice weekly for 12 weeks
  Arms: CP 690,550 10 mg BID+Placebo BIW
Biological: Etanercept 50 mg — Placebo orally dosed twice daily and etanercept 50 mg subcutaneously dosed twice weekly for 12 weeks
  Arms: Placebo BID+Etanercept 50 mg BIW
Other: Placebo — Placebo orally dosed twice daily and placebo subcutaneously dosed twice weekly for 12 weeks.
  Arms: Placebo BID+Placebo BIW

SUMMARY:
To evaluate the efficacy of CP-690,550 as compared to etanercept and the safety of CP-690,550 for treatment of moderate to severe chronic plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have had a diagnosis of plaque type psoriasis (psoriasis vulgaris);
* Have plaque-type psoriasis covering at least 10% of total body surface area
* Considered by dermatologist investigator to be a candidate for systemic therapy or phototherapy of psoriasis

Exclusion Criteria:

* Non-plaque or drug induced forms of psoriasis
* Cannot discontinue current systemic and/or topical therapies for the treatment of psoriasis
* Cannot discontinue phototherapy
* Any uncontrolled significant medical condition

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1101 (Actual)
Dates: Start 2010-11; Primary Completion 2013-01 (Actual); Study Completion 2013-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (122):
- Argentina (3):
  - Centro de Investigaciones Dermatologicas, Buenos Aires, C1114aap
  - Centro de Investigaciones Dermatologicas, Buenos Aires
  - IMAI (Instituto Medico de Asistencia e Investigaciones), Buenos Aires
- Austria (4):
  - LKH Feldkirch Abteilung fuer Dermatologie und Venerologie, Feldkirch
  - LKH Innsbruck Universitaetsklinik fuer Dermatologie und Venerologie, Innsbruck
  - LKH Salzburg, Landesklinik fuer Dermatologie, Salzburg
  - Krankenhaus Hietzing mit Neurologischem Zentrum Rosenhuegel, Vienna
- Belgium (2):
  - Cliniques universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
- Department for skin and venerial diseases, Clinical Center University of Sarajevo, Sarajevo, Bosnia and Herzegovina
- Bulgaria (5):
  - Universitetska Mnogoprofilna Bolnitsa Za Aktivno Lechenie- Dr Georgi Stranski- Pleven, Pleven
  - Tsentar za kozhno-venericheski zaboliavania" EOOD, Sofia
  - Mnogoprofilna Bolnitsa Za Aktivno Lechenie- Tokuda Bolnitsa Sofia- Sofia, Sofia
  - Universitetska mnogoprofilna bolnitsa za aktivno lechenie- Alexandrovska- Sofia, Sofia
  - MBAL na Voennomeditsinska akademia- Sofia, Sofia
- Chile (4):
  - Centro de Especialidades Dermatologicas, Viña del Mar, Región de Valparaíso
  - Clinica Davila, Santiago, Rm 8431657, RM
  - Clinica Dermovein S.A., Santiago
  - Hospital Clinico Universidad de Chile, Departamento Dermatologia, Santiago
- Colombia (5):
  - Reumalab S.A.S., Medellín, Antioquia
  - Centro Integral de Reumatología del Caribe Circaribe S.A, Barranquilla, Atlántico
  - Centro de Investigacion Clinica de la Universidad del Rosario, Bogota, Cundinamarca
  - Riesgo de Fractura S.A., Bogota, Cundinamarca
  - Medicity S.A.S, Bucaramanga, Santander Department
- Croatia (3):
  - Department of Dermatovenerology, University Hospital Center Osijek, Osijek
  - Dermatovenerological Clinic, University hospital center "Sestre milosrdnice", Zagreb
  - Department of dermatovenerology, University Hospital Center Zagreb, Zagreb
- Czechia (6):
  - Nemocnice Ceske Budejovice, a.s., České Budějovice
  - FN Kradec Kralove, Hradec Králové
  - Fakultni nemocnice Plzen, Plzen - Bory
  - Kozni ordinace, Prague
  - Kralska zdravotni a.s., Masarykovy nemocnice o.z., Ústí nad Labem
  - Kralska zdravotni, Ústí nad Labem
- Denmark (3):
  - Department of Dermatology, Aarhus University Hospital, Aarhus C
  - Bispebjerg Hospital, University of Copenhagen, Copenhagen NV
  - Hudklinikken Herning, Herning
- France (16):
  - CHG Le Mans, Le Mans, Cedex 09
  - CHU de Besancon - Hopital Saint Jacques, Besançon
  - Hopital Ambroise Pare, Service de Dermatologie, Boulogne
  - Chu Morvan, Brest Cédex
  - Hopital Dupuytren, Limoges
  - Hopital Fournier, Nancy Cédex
  - CHU de Nantes - Hotel Dieu, Nantes
  - CHU de NICE - Hôpital de l'Archet II, Nice
  - Hopital Saint-Louis, Paris
  - Hôpital Bichat, Paris
  - Centre Hospitalier Lyon Sud, Pierre-Bénite
  - C.H.U. de Poitiers, Poitiers
  - Hopital Robert Debre, Reims
  - Hopital Nord, Saint-Priest-en-Jarez
  - Hôpital Larrey, Toulouse
  - Hôpital de Brabois / Bâtiment Philippe Canton, Vandœuvre-lès-Nancy
- Germany (16):
  - Charite - Universitaetsmedizin Berlin, Berlin
  - Hautarztpraxis, Berlin
  - Dres.Kirsten Prepeneit und Volker Streit, Buchholz
  - Universitaets- Hautklinik Koeln, Cologne
  - Universitaetsklinik Carl Gustav Carus, Dresden
  - Hautzentrum Duelmen, Dülmen
  - Universitaetsklinikum Erlangen Hautklinik im Internistischen Zentrum, Erlangen
  - Klinikum der Johann Wolfgang Goethe Universitaet, Frankfurt am Main
  - Universitaetsklinikum Hamburg-Eppendorf, Hamburg
  - Hautklinik der Ruprecht-Karls-Universitaet Heidelberg, Heidelberg
  - Hautarztpraxis Dres. Scholz, Sebastian, Schilling, Mahlow
  - Universitaetsmedizin der Johannes Gutenberg-Universitaet Mainz KoeR, Mainz
  - Technische Universitaet Muenchen, München
  - Dres. med. Bredlich/PD Rosenbach/Thiele, Osnabrück
  - Eberhard-Karls-Universitaet Tuebingen, Tübingen
  - Hautarztpraxis, Witten
- The University of Hong Kong (HKU)-Queen Mary Hospital (QMH), Hong Kong, Hong Kong
- Hungary (5):
  - Synexus Magyarorszag Kft., Budapest
  - Debreceni Egyetem Orvos- es Egeszsegtudomanyi Centrum/Bor- es Nemikortani Klinika, Debrecen
  - Miskolci Semmelweis Ignac Korhaz-Rendelointezet/Borgyogyaszat, Miskolc
  - SZTE Szentgyorgyi Albert Klinikai Kozpont/Borgyogyaszati es Allergologiai Klinika, Szeged
  - ALLERGO-DERM BAKOS Kft., Szolnok
- Dermatology Department, Afula, Israel
- Netherlands (4):
  - Academic Medical Centre (AMC), Amsterdam, North Holland
  - PT & R, Beek
  - Amphia Hospital Location Molengracht / Department Dermatology, Breda
  - Erasmus MC, Rotterdam
- Poland (5):
  - NZOZ Osteo-Medic s.c. Artur Racewicz, Jerzy Supronik, Bialystok
  - Klinika Dermatologii, Wenerologii i Alergologii, Uniwersyteckie Centrum Kliniczne, Gdansk
  - Krakowskie Centrum Medyczne NZOZ, Krakow
  - Novum Instytut Dermatologii Leczniczej i Estetycznej, Opole
  - Solumed S.C., Poznan
- Russia (12):
  - Korolev Dermatovenerologic Dispensary, Korolyov, Moscow Oblast
  - State Research Center of Dermatovenerology, Department of clinical dermatology, Moscow
  - State Research Center of Dermatovenerology, Department of dermatology, Moscow
  - Dermatovenerologic dispensary #7, Moscow
  - Rostov-on-Don regional dermatovenerologic dispensary, Rostov-on-Don
  - Ryazan regional clinical dermatovenerologic dispensary, Ryazan
  - Dermatovenerologic dispensary #10 of Vyborg region, Saint Petersburg
  - Military medical academy S.M. Kirov, Saint Petersburg
  - North-Western State Medical University I.I. Mechnikov, Dermatovenerology Department, Saint Petersburg
  - Clinic of dermatovenerologic diseases, Saratov
  - Smolensk State Medical Academy, Smolensk
  - Clinical hospital of emergency care N.V. Soloviev, Yaroslavl
- Singapore (2):
  - National Skin Centre, Singapore
  - Changi General Hospital, Singapore
- Slovakia (3):
  - Dermatologicka klinika SZU, Fakultna nemocnica s poliklinikou F.D. Roosevelta, Banská Bystrica
  - Narodny ustav reumatickych chorob, Piešťany
  - DOST-Dermatovenerologicke oddelenie sanatorneho typu, SANARE, spol. s r.o., Svidník
- South Korea (2):
  - Samsung Medical Center / Department of Dermatology, Gangnam-Gu, Seoul
  - Severance Hospital, Yonsei University College of Medicine/Department of Dermatology, Seoul
- Spain (6):
  - Hospital Universitario Fundacion Alcorcon, Alcorcón, Madrid
  - Hospital Puerta de Hierro Majadahonda, Majadahonda, Madrid
  - Hospital General Universitario de Alicante, Alicante
  - Hospital Universitario de La Princesa, Madrid
  - Hospital 12 de Octubre, Madrid
  - Consorcio Hospital General Universitario de Valencia, Valencia
- Sweden (5):
  - Falu lasarett, Hudkliniken, Falun
  - Hermelinen Forskning AB, Luleå
  - Skanes Universitetssjukhus i Malmo, Hudkliniken, Malmo
  - Sodersjukhuset, Hudkliniken, Stockholm
  - Karolinska Universitetssjukhuset Solna, Stockholm
- Kantonsspital St. Gallen, Sankt Gallen, Switzerland
- Turkey (Türkiye) (5):
  - Gazi University Medical Faculty, Beşevler, Ankara
  - Istanbul university Istanbul Medical Faculty, Çapa, Istanbul
  - T.C. Saglik Bakanligi Marmara Universitesi Egitim ve Arastirma Hastanesi Dermatoloji Anabilim Dali, Pendik, Istanbul
  - Mersin University Medical Faculty, Akdeniz, Mersin
  - Dokuz Eylul Universitesi Tip Fakultesi Dermatoloji Anabilim Dali, Izmir
- United Kingdom (2):
  - Whipps Cross University Hospital, London, Leytonstone
  - Leicester Royal Infirmary, Balmoral building, Clinic 3, Dermatology, Leicester

REFERENCES:
- [Derived] Panaccione R, Isaacs JD, Chen LA, Wang W, Marren A, Kwok K, Wang L, Chan G, Su C. Characterization of Creatine Kinase Levels in Tofacitinib-Treated Patients with Ulcerative Colitis: Results from Clinical Trials. Dig Dis Sci. 2021 Aug;66(8):2732-2743. doi: 10.1007/s10620-020-06560-4. Epub 2020 Aug 20. PMID 32816215
- [Derived] Valenzuela F, Paul C, Mallbris L, Tan H, Papacharalambous J, Valdez H, Mamolo C. Tofacitinib versus etanercept or placebo in patients with moderate to severe chronic plaque psoriasis: patient-reported outcomes from a Phase 3 study. J Eur Acad Dermatol Venereol. 2016 Oct;30(10):1753-1759. doi: 10.1111/jdv.13702. Epub 2016 Jun 7. PMID 27271195
- [Derived] Bachelez H, van de Kerkhof PC, Strohal R, Kubanov A, Valenzuela F, Lee JH, Yakusevich V, Chimenti S, Papacharalambous J, Proulx J, Gupta P, Tan H, Tawadrous M, Valdez H, Wolk R; OPT Compare Investigators. Tofacitinib versus etanercept or placebo in moderate-to-severe chronic plaque psoriasis: a phase 3 randomised non-inferiority trial. Lancet. 2015 Aug 8;386(9993):552-61. doi: 10.1016/S0140-6736(14)62113-9. Epub 2015 Jun 4. PMID 26051365
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=A3921080&StudyName=A%20Phase%203%2C%20Multi%20Site%2C%20Randomized%2C%20Double%20Blind%2C%20Placebo%20Controlled%20Study%20Of%20The%20Efficacy%20And%20Safety%20Comparing%20CP-%20690%2C550%20And

RESULTS

PARTICIPANT FLOW:
Groups:
- CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW): Participants received CP-690,550 5 mg tablets, orally, BID, at approximately 12-hour intervals and placebo subcutaneous (SC) injections BIW at approximately 3- to 4-day intervals for 12 weeks.
- CP-690,550 10 mg BID + Placebo BIW: Participants received CP-690,550 10 mg tablets, orally, BID, at approximately 12-hour intervals and placebo SC injections BIW at approximately 3- to 4-day intervals for 12 weeks.
- Placebo BID + Etanercept 50 mg BIW: Participants received matching placebo tablets, orally, BID, at approximately 12-hour intervals and etanercept 50 mg SC injections BIW at approximately 3- to 4-day intervals for 12 weeks.
- Placebo BID + Placebo BIW: Participants received matching placebo tablets, orally, BID, at approximately 12-hour intervals and placebo SC injections BIW at approximately 3- to 4-day intervals for 12 weeks.
Period: Overall Study
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Started | 329 | 330 | 335 | 107
Completed | 306 | 306 | 313 | 95
Not Completed | 23 | 24 | 22 | 12
Not completed — Lack of Efficacy | 5 | 2 | 2 | 3
Not completed — Protocol Violation | 5 | 2 | 3 | 0
Not completed — Lost to Follow-up | 1 | 2 | 2 | 2
Not completed — Screen Failure | 3 | 2 | 1 | 0
Not completed — Withdrawal by Subject | 6 | 4 | 2 | 2
Not completed — Other | 0 | 1 | 0 | 1
Not completed — Adverse Event | 3 | 11 | 12 | 4

BASELINE CHARACTERISTICS:
Population: Full Analysis Set (FAS): included all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (CP-690,550, etanercept, or placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW | Total
Number analyzed (Participants) | 329 | 330 | 335 | 107 | 1101
Age, Continuous [Mean (Standard Deviation); unit: years] | 44.4 (12.1) | 43.6 (12.6) | 43.3 (12.2) | 46.1 (13.4) | 44.0 (12.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 93 | 92 | 102 | 36 | 323
  Male | 236 | 238 | 233 | 71 | 778

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants With a Physician's Global Assessment (PGA) Response of "Clear" or "Almost Clear" at Week 12
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 to 4). The severity scores are summed and averaged after which the total average is rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response was defined as 0 (clear) or 1 (almost clear).
Time Frame: Week 12
Population: Full Analysis Set (FAS): all participants who were randomized to the study and received at least 1 dose of the randomized investigational drug (CP-690,550, etanercept, or placebo); Non-Responder Imputation (NRI) method: participants with missing values were considered to be non-responders.
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 329 | 330 | 335 | 107
percentage of participants | 47.11 | 68.18 | 66.27 | 14.95
Statistical Analysis 1: Comparison: CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) vs Placebo BID + Etanercept 50 mg BIW; Difference from Etanercept (Active-Etanercept); Test type: Non-Inferiority or Equivalence — The a priori threshold for non-inferiority was -15% and a step-down approach was used to adjust for multiple comparisons. Non-inferiority of CP-690,550 5 mg to etanercept was concluded if the 95% lower confidence intervals (LCIs) of the difference for PGA and Psoriasis Area and Severity Index 75 (PASI75) responses at Week 12 were greater than -15%, and CP-690,550 10 mg was superior to placebo for PGA response and PASI75 at Week 12; Mean Difference = -19.16, 95% CI 2-sided [-26.55 to -11.76], Standard Error of Mean 3.77
Statistical Analysis 2: Comparison: CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) vs Placebo BID + Placebo BIW; Difference from Placebo (Active-Placebo); the a priori threshold for superiority was 0 and a step-down approach was used to adjust for multiple comparisons. Superiority of CP-690,550 5 mg to placebo was concluded if the lower bounds of the 95% LCIs of the difference for PGA and PASI75 responses at Week 12 were greater than 0, and non-inferiority of CP-690,550 5 mg was concluded to be non-inferior to etanercept; Test type: Superiority or Other; Mean Difference = 32.16, 95% CI 2-sided [23.51 to 40.81], Standard Error of Mean 4.41
Statistical Analysis 3: Comparison: CP-690,550 10 mg BID + Placebo BIW vs Placebo BID + Etanercept 50 mg BIW; Difference from Etanercept (Active-Etanercept); Test type: Non-Inferiority or Equivalence — The a priori threshold for non-inferiority was -15% and a step-down approach was used to adjust for multiple comparisons. Non-inferiority of CP-690,550 10 mg to etanercept was concluded if the 95% LCIs of the difference for PGA and PASI75 responses at Week 12 were greater than -15%; Mean Difference = 1.91, 95% CI 2-sided [-5.22 to 9.05], Standard Error of Mean 3.64
Statistical Analysis 4: Comparison: CP-690,550 10 mg BID + Placebo BIW vs Placebo BID + Placebo BIW; Difference from Placebo (Active-Placebo); the a priori threshold for superiority was 0 and a step-down approach was used to adjust for multiple comparisons. Superiority of CP-690,550 10 mg to placebo was concluded if the 95% LCIs of the difference for PGA and PASI75 responses at Week 12 were greater than 0, and non-inferiority of CP-690,550 10 mg was concluded to be non-inferior to etanercept; Test type: Superiority or Other; Mean Difference = 53.23, 95% CI 2-sided [44.81 to 61.65], Standard Error of Mean 4.30

2. Primary Outcome: Percentage of Participants With a Psoriasis Area and Severity Index 75 (PASI75) Response at Week 12
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percent of body surface area (BSA) affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI75 response was defined as at least a 75 percent (%) reduction in PASI relative to baseline/Day 1.
Time Frame: Week 12
Population: FAS; NRI
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 329 | 330 | 335 | 107
percentage of participants | 39.51 | 63.64 | 58.81 | 5.61
Statistical Analysis 1: Comparison: CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) vs Placebo BID + Etanercept 50 mg BIW; Difference from Etanercept (Active-Etanercept); Test type: Non-Inferiority or Equivalence — The a priori threshold for non-inferiority was -15% and a step-down approach was used to adjust for multiple comparisons. Non-inferiority of CP-690,550 5 mg to etanercept was concluded if the 95% LCIs of the difference for PGA and PASI75 responses at Week 12 were greater than -15%, and CP-690,550 10 mg was superior to placebo for PGA and PASI75 response at Week 12; Mean Difference = -19.29, 95% CI 2-sided [-26.75 to -11.83], Standard Error of Mean 3.81
Statistical Analysis 2: Comparison: CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) vs Placebo BID + Placebo BIW; Difference from Placebo (Active-Placebo); the a priori threshold for superiority was 0 and a step-down approach was used to adjust for multiple comparisons. Superiority of CP-690,550 5 mg to placebo was concluded if the 95% LCIs of the difference for PGA and PASI75 responses at Week 12 were greater than 0, and non-inferiority of CP-690,550 5 mg was concluded to be non-inferior to etanercept; Test type: Superiority or Other; Mean Difference = 33.91, 95% CI 2-sided [27.06 to 40.76], Standard Error of Mean 3.49
Statistical Analysis 3: Comparison: CP-690,550 10 mg BID + Placebo BIW vs Placebo BID + Etanercept 50 mg BIW; Difference from Etanercept (Active-Etanercept); Test type: Non-Inferiority or Equivalence — [test comment as in outcome 1, analysis 3]; Mean Difference = 4.83, 95% CI 2-sided [-2.57 to 12.23], Standard Error of Mean 3.77
Statistical Analysis 4: Comparison: CP-690,550 10 mg BID + Placebo BIW vs Placebo BID + Placebo BIW; [analysis description as in outcome 1, analysis 4]; Test type: Superiority or Other; Mean Difference = 58.03, 95% CI 2-sided [51.25 to 64.81], Standard Error of Mean 3.46

3. Secondary Outcome: Percentage of Participants With a PGA Response of "Clear" or "Almost Clear" During the 12-Week Double-Blind Treatment
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 to 4). The severity scores are summed and averaged after which the total average is rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe). PGA response is defined as 0 (clear) or 1 (almost clear).
Time Frame: Weeks 2, 4, and 8
Population: FAS; Observed Case (OC): no imputation
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 325 | 326 | 331 | 107
percentage of participants
  Week 2 (n=325,326,331,107) | 6.77 | 10.74 | 7.85 | 1.87
  Week 4 (n=320,323,328,102) | 21.25 | 35.91 | 28.35 | 3.92
  Week 8 (n=314,316,322,100) | 40.45 | 63.61 | 60.87 | 13.00

4. Secondary Outcome: Percentage of Participants in Each PGA Category During the 12-Week Double-Blind Treatment
Description: The PGA of psoriasis is scored on a 5-point scale, reflecting a global consideration of the erythema, induration, and scaling across all psoriatic lesions. Average erythema, induration, and scaling are scored separately over the whole body according to a 5-point severity scale (0 to 4). The severity scores are summed and averaged after which the total average is rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe).
Time Frame: Baseline and Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 329 | 330 | 335 | 107
percentage of participants
  Baseline, Clear (n=329,330,335,107) | 0.0 | 0.0 | 0.0 | 0.0
  Baseline, Almost Clear (n=329,330,335,107) | 0.0 | 0.0 | 0.0 | 0.0
  Baseline, Mild (n=329,330,335,107) | 1.8 | 1.2 | 1.2 | 2.8
  Baseline, Moderate (n=329,330,335,107) | 80.2 | 83.3 | 80.9 | 82.2
  Baseline, Severe (n=329,330,335,107) | 17.9 | 15.5 | 17.9 | 15.0
  Week 2, Clear (n=325,326,331,107) | 0.0 | 0.0 | 0.0 | 0.0
  Week 2, Almost Clear (n=325,326,331,107) | 6.8 | 10.7 | 7.9 | 1.9
  Week 2, Mild (n=325,326,331,107) | 38.5 | 47.9 | 42.6 | 25.2
  Week 2, Moderate (n=325,326,331,107) | 48.9 | 38.3 | 45.6 | 64.5
  Week 2, Severe (n=325,326,331,107) | 5.8 | 3.1 | 3.9 | 8.4
  Week 4, Clear (n=320,323,328,102) | 1.9 | 2.5 | 0.6 | 0.0
  Week 4, Almost Clear (n=320,323,328,102) | 19.4 | 33.4 | 27.7 | 3.9
  Week 4, Mild (n=320,323,328,102) | 46.3 | 44.3 | 51.5 | 34.3
  Week 4, Moderate (n=320,323,328,102) | 30.0 | 17.6 | 19.5 | 55.9
  Week 4, Severe (n=320,323,328,102) | 2.5 | 2.2 | 0.6 | 5.9
  Week 8, Clear (n=314,316,322,100) | 5.4 | 14.2 | 9.0 | 0.0
  Week 8, Almost Clear (n=314,316,322,100) | 35.0 | 49.4 | 51.9 | 13.0
  Week 8, Mild (n=314,316,322,100) | 41.4 | 25.0 | 30.1 | 35.0
  Week 8, Moderate (n=314,316,322,100) | 15.9 | 10.8 | 8.1 | 49.0
  Week 8, Severe (n=314,316,322,100) | 2.2 | 0.6 | 0.9 | 3.0
  Week 12, Clear (n=314,316,322,100) | 11.8 | 27.0 | 21.0 | 2.1
  Week 12, Almost Clear (n=313,311,309,95) | 37.7 | 45.3 | 50.8 | 14.7
  Week 12, Mild (n=313,311,309,95) | 33.5 | 19.3 | 21.4 | 36.8
  Week 12, Moderate (n=313,311,309,95) | 15.7 | 7.4 | 5.5 | 42.1
  Week 12, Severe (n=313,311,309,95) | 1.3 | 1.0 | 1.3 | 4.2

5. Secondary Outcome: Percentage of Participants With a PASI75 Response During the 12-Week Double-Blind Treatment
Description: The PASI quantifies the severity of a participant's psoriasis based on both lesion severity and the percent of BSA affected. PASI is a composite scoring by the investigator of degree of erythema, induration, and scaling (each scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0, with higher scores representing greater severity of psoriasis. PASI75 response was defined as at least a 75% reduction in PASI relative to baseline/Day 1.
Time Frame: Weeks 2, 4, and 8
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 326 | 327 | 331 | 106
percentage of participants
  Week 2 (n=326,327,331,106) | 1.53 | 2.75 | 0.91 | 0.00
  Week 4 (n=319,323,328,102) | 10.34 | 19.81 | 8.23 | 0.00
  Week 8 (n=315,319,323,99) | 28.57 | 52.35 | 42.72 | 3.03

6. Secondary Outcome: Mean PASI Score During the 12-Week Double-Blind Treatment
Description: Combined assessment of lesion severity and area affected into single score; range=0(no disease)-72(maximal disease). Body divided into 4 sections=head, upper/lower limbs, trunk; each area scored by itself and scores combined for final PASI. For each section percent area of skin involved was estimated:0(0%)-6(90-100%) and severity estimated by clinical signs of erythema, induration, scaling; ranged 0-4: 0=none, 1=slight, 2=moderate, 3=marked, 4=very marked. Final PASI=sum of severity parameters for each section*area score*weighing factor (head=0.1, upper limbs=0.2, trunk=0.3, lower limbs=0.4). PASI score can vary in increments of 0.1; higher scores represent greater severity of psoriasis.
Time Frame: Baseline and Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 329 | 330 | 335 | 107
score on a scale
  Baseline (n=329,330,335,107) | 23.13 (0.48) | 23.29 (0.53) | 22.73 (0.53) | 22.78 (0.88)
  Week 2 (n=326,327,328,102) | 18.16 (0.47) | 16.81 (0.53) | 17.29 (0.49) | 21.26 (0.95)
  Week 4 (n=319,323,328,102) | 14.46 (0.46) | 12.13 (0.52) | 12.73 (0.44) | 20.06 (0.94)
  Week 8 (n=315,319,323,99) | 10.63 (0.44) | 7.59 (0.48) | 7.70 (0.38) | 17.91 (0.99)
  Week 12 (n=313,311,309,95) | 8.80 (0.43) | 5.77 (0.45) | 5.42 (0.36) | 17.39 (1.06)

7. Secondary Outcome: Mean Change From Baseline in PASI Score During the 12-Week Double-Blind Treatment
Description: as for outcome 6
Time Frame: Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 326 | 327 | 331 | 106
scores on a scale
  Week 2 (n=326,327,331,106) | -5.03 (0.31) | -6.47 (0.31) | -5.48 (0.29) | -1.58 (0.46)
  Week 4 (n=319,323,328,102) | -8.83 (0.42) | -11.30 (0.43) | -10.14 (0.39) | -2.58 (0.62)
  Week 8 (n=315,319,323,99) | -12.62 (0.52) | -15.81 (0.51) | -15.20 (0.51) | -4.82 (0.81)
  Week 12 (n=313,311,309,95) | -14.55 (0.60) | -17.54 (0.54) | -17.55 (0.57) | -5.33 (0.97)

8. Secondary Outcome: Mean PASI Component Scores by Body Region During the 12-Week Double Blind Treatment
Description: as for outcome 6
Time Frame: Baseline and Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 329 | 329 | 335 | 107
score on a scale
  Head/Neck Erythema, Baseline (n=329,329,335,107) | 2.28 (0.05) | 2.36 (0.05) | 2.32 (0.05) | 2.40 (0.09)
  Head/Neck Erythema, Week 2 (n=326,326,331,106) | 1.82 (0.05) | 1.65 (0.05) | 1.76 (0.06) | 2.27 (0.09)
  Head/Neck Erythema, Week 4 (n=320,323,328,102) | 1.48 (0.05) | 1.18 (0.05) | 1.23 (0.05) | 2.03 (0.09)
  Head/Neck Erythema, Week 8 (n=315,319,323,99) | 1.19 (0.06) | 0.78 (0.05) | 0.69 (0.05) | 1.89 (0.10)
  Head/Neck Erythema, Week 12 (n=313,311,309,95) | 1.04 (0.06) | 0.65 (0.05) | 0.48 (0.04) | 1.74 (0.11)
  Head/Neck Induration, Baseline (n=329,329,335,107) | 2.04 (0.05) | 2.08 (0.05) | 1.96 (0.06) | 2.12 (0.10)
  Head/Neck Induration, Week 2 (n=326,326,331,106) | 1.60 (0.05) | 1.44 (0.05) | 1.46 (0.06) | 1.97 (0.10)
  Head/Neck Induration, Week 4 (n=320,323,328,102) | 1.21 (0.05) | 0.94 (0.05) | 1.01 (0.05) | 1.69 (0.10)
  Head/Neck Induration, Week 8 (n=315,319,323,99) | 0.96 (0.05) | 0.59 (0.05) | 0.54 (0.05) | 1.57 (0.10)
  Head/Neck Induration, Week 12 (n=313,311,309,95) | 0.87 (0.05) | 0.49 (0.04) | 0.37 (0.04) | 1.41 (0.11)
  Head/Neck Scaling, Baseline (n=329,329,335,107) | 2.29 (0.06) | 2.38 (0.06) | 2.28 (0.06) | 2.33 (0.10)
  Head/Neck Scaling, Week 2 (n=326,326,331,106) | 1.75 (0.06) | 1.63 (0.06) | 1.60 (0.06) | 2.15 (0.10)
  Head/Neck Scaling, Week 4 (n=320,323,328,102) | 1.38 (0.06) | 1.07 (0.06) | 1.16 (0.05) | 1.80 (0.11)
  Head/Neck Scaling, Week 8 (n=315,319,323,99) | 1.12 (0.06) | 0.70 (0.05) | 0.65 (0.05) | 1.66 (0.11)
  Head/Neck Scaling, Week 12 (n=313,311,309,95) | 0.98 (0.06) | 0.60 (0.05) | 0.46 (0.05) | 1.51 (0.11)
  Upper Limbs Erythema, Baseline (n=329,329,335,107) | 2.87 (0.04) | 2.87 (0.04) | 2.88 (0.04) | 2.92 (0.07)
  Upper Limbs Erythema, Week 2 (n=326,326,331,106) | 2.35 (0.04) | 2.18 (0.05) | 2.27 (0.05) | 2.75 (0.07)
  Upper Limbs Erythema, Week 4 (n=320,323,328,102) | 1.92 (0.05) | 1.73 (0.05) | 1.77 (0.05) | 2.61 (0.07)
  Upper Limbs Erythema, Week 8 (n=315,319,323,99) | 1.55 (0.05) | 1.27 (0.05) | 1.25 (0.05) | 2.42 (0.08)
  Upper Limbs Erythema, Week 12 (n=313,311,309,95) | 1.45 (0.06) | 1.07 (0.05) | 0.94 (0.05) | 2.32 (0.08)
  Upper Limbs Induration Baseline(n=329,329,335,107) | 2.69 (0.04) | 2.76 (0.04) | 2.72 (0.04) | 2.79 (0.07)
  Upper Limbs Induration, Week 2 (n=326,326,331,106) | 2.17 (0.05) | 2.03 (0.05) | 2.13 (0.05) | 2.54 (0.07)
  Upper Limbs Induration, Week 4 (n=320,323,328,102) | 1.76 (0.05) | 1.54 (0.05) | 1.59 (0.05) | 2.36 (0.08)
  Upper Limbs Induration, Week 8 (n=315,319,323,99) | 1.43 (0.06) | 1.13 (0.05) | 1.18 (0.05) | 2.12 (0.09)
  Upper Limbs Induration, Week 12 (n=313,311,309,95) | 1.31 (0.06) | 1.01 (0.05) | 0.81 (0.05) | 2.08 (0.09)
  Upper Limbs Scaling, Baseline (n=329,329,335,107) | 2.66 (0.04) | 2.72 (0.04) | 2.73 (0.04) | 2.63 (0.08)
  Upper Limbs Scaling, Week 2 (n=326,326,331,106) | 2.11 (0.05) | 2.00 (0.05) | 2.03 (0.05) | 2.35 (0.09)
  Upper Limbs Scaling, Week 4 (n=320,323,328,102) | 1.71 (0.05) | 1.50 (0.05) | 1.54 (0.05) | 2.22 (0.10)
  Upper Limbs Scaling, Week 8 (n=315,319,323,99) | 1.39 (0.06) | 1.11 (0.05) | 1.07 (0.05) | 1.98 (0.09)
  Upper Limbs Scaling, Week 12 (n=313,311,309,95) | 1.30 (0.06) | 1.00 (0.05) | 0.82 (0.05) | 1.95 (0.10)
  Trunk Erythema, Baseline (n=329,329,335,107) | 2.95 (0.04) | 2.88 (0.04) | 2.91 (0.04) | 2.97 (0.06)
  Trunk Erythema, Week 2 (n=326,326,331,106) | 2.40 (0.05) | 2.20 (0.05) | 2.27 (0.05) | 2.75 (0.07)
  Trunk Erythema, Week 4 (n=320,323,328,102) | 2.03 (0.05) | 1.75 (0.05) | 1.76 (0.05) | 2.59 (0.07)
  Trunk Erythema, Week 8 (n=315,319,323,99) | 1.71 (0.06) | 1.23 (0.05) | 1.24 (0.05) | 2.41 (0.09)
  Trunk Erythema, Week 12 (n=313,311,309,95) | 1.53 (0.06) | 0.97 (0.06) | 0.89 (0.05) | 2.33 (0.10)
  Trunk Induration, Baseline (n=329,329,335,107) | 2.75 (0.04) | 2.70 (0.05) | 2.66 (0.05) | 2.66 (0.07)
  Trunk Induration, Week 2 (n=326,326,331,106) | 2.26 (0.05) | 2.01 (0.05) | 2.05 (0.05) | 2.40 (0.07)
  Trunk Induration, Week 4 (n=320,323,328,102) | 1.83 (0.05) | 1.50 (0.05) | 1.50 (0.05) | 2.26 (0.07)
  Trunk Induration, Week 8 (n=315,319,323,99) | 1.50 (0.06) | 0.97 (0.05) | 0.98 (0.05) | 2.06 (0.09)
  Trunk Induration, Week 12 (n=313,311,309,95) | 1.33 (0.06) | 0.80 (0.05) | 0.66 (0.05) | 2.03 (0.09)
  Trunk Scaling, Baseline (n=329,329,335,107) | 2.64 (0.04) | 2.66 (0.05) | 2.57 (0.05) | 2.61 (0.07)
  Trunk Scaling, Week 2 (n=326,326,331,106) | 2.12 (0.05) | 1.92 (0.06) | 1.93 (0.05) | 2.36 (0.09)
  Trunk Scaling, Week 4 (n=320,323,328,102) | 1.73 (0.05) | 1.39 (0.05) | 1.44 (0.05) | 2.12 (0.09)
  Trunk Scaling, Week 8 (n=315,319,323,99) | 1.47 (0.06) | 0.94 (0.05) | 0.90 (0.05) | 1.86 (0.08)
  Trunk Scaling, Week 12 (n=313,311,309,95) | 1.28 (0.06) | 0.74 (0.05) | 0.62 (0.05) | 1.91 (0.10)
  Lower Limbs Erythema, Baseline (n=329,329,335,107) | 3.12 (0.03) | 3.13 (0.04) | 3.14 (0.03) | 3.10 (0.06)
  Lower Limbs Erythema, Week 2 (n=326,326,331,106) | 2.60 (0.04) | 2.44 (0.05) | 2.61 (0.05) | 2.92 (0.07)
  Lower Limbs Erythema, Week 4 (n=320,323,328,102) | 2.17 (0.05) | 1.98 (0.05) | 2.15 (0.05) | 2.75 (0.07)
  Lower Limbs Erythema, Week 8 (n=315,319,323,99) | 1.77 (0.06) | 1.50 (0.05) | 1.62 (0.05) | 2.55 (0.08)
  Lower Limbs Erythema, Week 12 (n=313,311,309,95) | 1.56 (0.06) | 1.21 (0.06) | 1.35 (0.05) | 2.45 (0.09)
  Lower Limbs Induration Baseline(n=329,329,335,107) | 2.94 (0.04) | 2.97 (0.04) | 3.00 (0.04) | 2.92 (0.07)
  Lower Limbs Induration, Week 2 (n=326,326,331,106) | 2.47 (0.04) | 2.26 (0.05) | 2.45 (0.04) | 2.69 (0.07)
  Lower Limbs Induration, Week 4 (n=320,323,328,102) | 2.03 (0.05) | 1.72 (0.05) | 1.92 (0.05) | 2.54 (0.07)
  Lower Limbs Induration, Week 8 (n=315,319,323,99) | 1.58 (0.06) | 1.18 (0.05) | 1.38 (0.05) | 2.25 (0.08)
  Lower Limbs Induration, Week 12 (n=313,311,309,95) | 1.40 (0.06) | 0.97 (0.05) | 1.10 (0.06) | 2.21 (0.08)
  Lower Limbs Scaling, Baseline (n=329,329,335,107) | 2.91 (0.04) | 2.95 (0.04) | 2.98 (0.04) | 2.89 (0.07)
  Lower Limbs Scaling, Week 2 (n=326,326,331,106) | 2.36 (0.05) | 2.25 (0.05) | 2.31 (0.05) | 2.62 (0.09)
  Lower Limbs Scaling, Week 4 (n=320,323,328,102) | 1.98 (0.05) | 1.69 (0.06) | 1.81 (0.05) | 2.44 (0.09)
  Lower Limbs Scaling, Week 8 (n=315,319,323,99) | 1.60 (0.06) | 1.21 (0.06) | 1.32 (0.05) | 2.11 (0.10)
  Lower Limbs Scaling, Week 12 (n=313,311,309,95) | 1.39 (0.06) | 0.96 (0.06) | 1.08 (0.06) | 2.09 (0.10)

9. Secondary Outcome: Mean Change From Baseline in PASI Component Scores by Body Region During the 12-Week Double Blind Treatment
Description: as for outcome 6
Time Frame: Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 326 | 326 | 331 | 106
scores on a scale
  Head/Neck Erythema, Week 2 (n=326,326,331,106) | -0.46 (0.04) | -0.72 (0.05) | -0.56 (0.04) | -0.15 (0.06)
  Head/Neck Erythema, Week 4 (n=320,323,328,102) | -0.80 (0.06) | -1.19 (0.06) | -1.10 (0.05) | -0.32 (0.07)
  Head/Neck Erythema, Week 8 (n=315,319,323,99) | -1.09 (0.06) | -1.59 (0.06) | -1.63 (0.06) | -0.54 (0.10)
  Head/Neck Erythema, Week 12 (n=313,311,309,95) | -1.25 (0.07) | -1.73 (0.07) | -1.83 (0.06) | -0.64 (0.12)
  Head/Neck Induration, Week 2 (n=326,326,331,106) | -0.44 (0.04) | -0.65 (0.05) | -0.49 (0.04) | -0.17 (0.06)
  Head/Neck Induration, Week 4 (n=320,323,328,102) | -0.83 (0.06) | -1.15 (0.06) | -0.95 (0.05) | -0.39 (0.08)
  Head/Neck Induration, Week 8 (n=315,319,323,99) | -1.08 (0.06) | -1.50 (0.06) | -1.41 (0.06) | -0.58 (0.10)
  Head/Neck Induration, Week 12 (n=313,311,309,95) | -1.19 (0.06) | -1.61 (0.06) | -1.57 (0.06) | -0.71 (0.11)
  Head/Neck Scaling, Week 2 (n=326,326,331,106) | -0.53 (0.04) | -0.76 (0.05) | -0.67 (0.05) | -0.20 (0.07)
  Head/Neck Scaling, Week 4 (n=320,323,328,102) | -0.91 (0.06) | -1.30 (0.07) | -1.13 (0.06) | -0.48 (0.08)
  Head/Neck Scaling, Week 8 (n=315,319,323,99) | -1.16 (0.07) | -1.70 (0.06) | -1.62 (0.06) | -0.69 (0.10)
  Head/Neck Scaling, Week 12 (n=313,311,309,95) | -1.31 (0.07) | -1.78 (0.07) | -1.81 (0.07) | -0.80 (0.11)
  Upper Limbs Erythema, Week 2 (n=326,326,331,106) | -0.52 (0.04) | -0.68 (0.04) | -0.61 (0.04) | -0.18 (0.06)
  Upper Limbs Erythema, Week 4 (n=320,323,328,102) | -0.94 (0.05) | -1.13 (0.05) | -1.11 (0.04) | -0.26 (0.07)
  Upper Limbs Erythema, Week 8 (n=315,319,323,99) | -1.31 (0.06) | -1.60 (0.06) | -1.62 (0.05) | -0.49 (0.08)
  Upper Limbs Erythema, Week 12 (n=313,311,309,95) | -1.42 (0.07) | -1.79 (0.06) | -1.95 (0.06) | -0.58 (0.09)
  Upper Limbs Induration, Week 2 (n=326,326,331,106) | -0.52 (0.04) | -0.73 (0.04) | -0.59 (0.04) | -0.25 (0.05)
  Upper Limbs Induration, Week 4 (n=320,323,328,102) | -0.94 (0.06) | -1.23 (0.05) | -1.13 (0.05) | -0.39 (0.07)
  Upper Limbs Induration, Week 8 (n=315,319,323,99) | -1.26 (0.06) | -1.65 (0.06) | -1.54 (0.05) | -0.67 (0.08)
  Upper Limbs Induration, Week 12 (n=313,311,309,95) | -1.39 (0.07) | -1.77 (0.06) | -1.92 (0.06) | -0.68 (0.10)
  Upper Limbs Scaling, Week 2 (n=326,326,331,106) | -0.56 (0.04) | -0.72 (0.05) | -0.69 (0.04) | -0.28 (0.07)
  Upper Limbs Scaling, Week 4 (n=320,323,328,102) | -0.96 (0.05) | -1.23 (0.06) | -1.19 (0.05) | -0.38 (0.08)
  Upper Limbs Scaling, Week 8 (n=315,319,323,99) | -1.28 (0.06) | -1.62 (0.06) | -1.66 (0.06) | -0.64 (0.08)
  Upper Limbs Scaling, Week 12 (n=313,311,309,95) | -1.36 (0.07) | -1.73 (0.06) | -1.92 (0.06) | -0.65 (0.10)
  Trunk Erythema, Week 2 (n=326,326,331,106) | -0.54 (0.04) | -0.67 (0.04) | -0.63 (0.04) | -0.23 (0.06)
  Trunk Erythema, Week 4 (n=320,323,328,102) | -0.91 (0.05) | -1.13 (0.05) | -1.16 (0.05) | -0.35 (0.06)
  Trunk Erythema, Week 8 (n=315,319,323,99) | -1.23 (0.06) | -1.66 (0.06) | -1.67 (0.06) | -0.59 (0.08)
  Trunk Erythema, Week 12 (n=313,311,309,95) | -1.41 (0.07) | -1.90 (0.07) | -2.03 (0.06) | -0.67 (0.10)
  Trunk Induration, Week 2 (n=326,326,331,106) | -0.49 (0.04) | -0.69 (0.04) | -0.61 (0.04) | -0.27 (0.06)
  Trunk Induration, Week 4 (n=320,323,328,102) | -0.93 (0.06) | -1.20 (0.06) | -1.17 (0.05) | -0.37 (0.07)
  Trunk Induration, Week 8 (n=315,319,323,99) | -1.26 (0.06) | -1.74 (0.06) | -1.68 (0.06) | -0.62 (0.10)
  Trunk Induration, Week 12 (n=313,311,309,95) | -1.43 (0.07) | -1.91 (0.07) | -1.99 (0.06) | -0.64 (0.11)
  Trunk Scaling, Week 2 (n=326,326,331,106) | -0.52 (0.05) | -0.74 (0.05) | -0.64 (0.05) | -0.25 (0.07)
  Trunk Scaling, Week 4 (n=320,323,328,102) | -0.92 (0.06) | -1.27 (0.06) | -1.15 (0.05) | -0.47 (0.08)
  Trunk Scaling, Week 8 (n=315,319,323,99) | -1.19 (0.06) | -1.71 (0.06) | -1.67 (0.06) | -0.75 (0.09)
  Trunk Scaling, Week 12 (n=313,311,309,95) | -1.38 (0.07) | -1.92 (0.06) | -1.94 (0.06) | -0.71 (0.10)
  Lower Limbs Erythema, Week 2 (n=326,326,331,106) | -0.52 (0.04) | -0.69 (0.04) | -0.53 (0.04) | -0.20 (0.05)
  Lower Limbs Erythema, Week 4 (n=320,323,328,102) | -0.95 (0.05) | -1.15 (0.05) | -1.00 (0.04) | -0.32 (0.06)
  Lower Limbs Erythema, Week 8 (n=315,319,323,99) | -1.34 (0.06) | -1.63 (0.05) | -1.51 (0.05) | -0.55 (0.08)
  Lower Limbs Erythema, Week 12 (n=313,311,309,95) | -1.55 (0.07) | -1.92 (0.07) | -1.80 (0.06) | -0.61 (0.09)
  Lower Limbs Induration, Week 2 (n=326,326,331,106) | -0.47 (0.04) | -0.71 (0.04) | -0.56 (0.04) | -0.24 (0.05)
  Lower Limbs Induration, Week 4 (n=320,323,328,102) | -0.92 (0.05) | -1.25 (0.05) | -1.08 (0.05) | -0.35 (0.07)
  Lower Limbs Induration, Week 8 (n=315,319,323,99) | -1.37 (0.06) | -1.80 (0.06) | -1.62 (0.06) | -0.66 (0.08)
  Lower Limbs Induration, Week 12 (n=313,311,309,95) | -1.56 (0.07) | -2.01 (0.06) | -1.91 (0.06) | -0.67 (0.09)
  Lower Limbs Scaling, Week 2 (n=326,326,331,106) | -0.55 (0.04) | -0.69 (0.05) | -0.67 (0.04) | -0.27 (0.06)
  Lower Limbs Scaling, Week 4 (n=320,323,328,102) | -0.94 (0.05) | -1.26 (0.06) | -1.18 (0.05) | -0.43 (0.09)
  Lower Limbs Scaling, Week 8 (n=315,319,323,99) | -1.31 (0.06) | -1.74 (0.06) | -1.67 (0.06) | -0.75 (0.09)
  Lower Limbs Scaling, Week 12 (n=313,311,309,95) | -1.53 (0.07) | -1.99 (0.06) | -1.92 (0.07) | -0.76 (0.10)

10. Secondary Outcome: Mean Percentage of Total Psoriatic BSA During the 12-Week Double-Blind Treatment
Description: Assessment of BSA with psoriasis performed separately for 4 body regions: head and neck, upper limbs, trunk (including axillae and groin), and lower limbs (including buttocks). The % surface area with psoriasis was estimated by means of the handprint method, where the full palmar hand of the participant (fully extended palm, fingers and thumb together) represented approximately 1% of the total BSA. The number of handprints of psoriatic skin in a body region was used to determine the extent (%) to which a body region was involved with psoriasis.
Time Frame: Baseline and Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: percent psoriatic BSA
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 329 | 329 | 335 | 107
percent psoriatic BSA
  Baseline (n=329,329,335,107) | 32.15 (0.98) | 31.74 (0.95) | 30.63 (1.00) | 31.88 (1.62)
  Week 2 (n=326,326,331,106) | 29.53 (0.96) | 28.12 (0.94) | 28.29 (0.97) | 32.03 (1.76)
  Week 4 (n=320,323,328,102) | 25.98 (0.96) | 22.88 (0.93) | 24.82 (0.95) | 32.47 (1.89)
  Week 8 (n=315,319,323,99) | 19.74 (0.98) | 14.76 (0.89) | 15.42 (0.81) | 31.00 (1.98)
  Week 12 (n=313,311,309,95) | 16.04 (0.94) | 10.55 (0.77) | 10.60 (0.76) | 29.77 (2.12)

11. Secondary Outcome: Mean Percent Change From Baseline in Total Psoriatic BSA During the 12-Week Double-Blind Treatment
Description: Assessment of BSA with psoriasis performed separately for 4 body regions: head and neck, upper limbs, trunk (including axillae and groin), and lower limbs (including buttocks). The %surface area with psoriasis was estimated by means of the handprint method, where the full palmar hand of the participant(fully extended palm, fingers and thumb together) represented approximately 1% of the total BSA. The number of handprints of psoriatic skin in a body region was used to determine the extent (%) to which a body region was involved with psoriasis.
Time Frame: Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: percent change from baseline
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 326 | 326 | 331 | 106
percent change from baseline
  Week 2 (n=326,326,331,106) | -7.54 (1.23) | -11.71 (1.12) | -7.54 (0.96) | 0.23 (1.89)
  Week 4 (n=320,323,328,102) | -19.90 (1.66) | -29.17 (1.69) | -19.60 (1.46) | 1.58 (2.84)
  Week 8 (n=315,319,323,99) | -37.81 (2.81) | -55.02 (1.93) | -48.65 (1.91) | -1.33 (3.57)
  Week 12 (n=313,311,309,95) | -47.66 (3.35) | -67.51 (1.86) | -64.91 (1.91) | -6.68 (4.06)

12. Secondary Outcome: Percentage of Participants Who Achieved a 50% Reduction in PASI Relative to Baseline (PASI50) During the 12-Week Double-Blind Treatment
Description: PASI quantifies severity of psoriasis based on both lesion severity and percent of BSA affected. PASI is a composite score by the investigator of degree of erythema, induration, and scaling (scored separately) for each of 4 body regions (head and neck, upper limbs, trunk [including axillae and groin], and lower limbs [including buttocks), with adjustment for the percent of BSA involved for each body region and for the proportion of the body region to the whole body. The PASI score can vary in increments of 0.1 and range from 0.0 to 72.0; higher scores represent greater severity of psoriasis.
Time Frame: Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Number; unit: percentage of participatns
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 326 | 327 | 331 | 106
percentage of participatns
  Week 2 (n=326,327,331,106) | 10.74 | 18.35 | 11.18 | 0.94
  Week 4 (n=319,323,328,102) | 33.23 | 50.46 | 48.78 | 6.86
  Week 8 (n=315,319, 323,99) | 59.05 | 78.06 | 77.09 | 20.20
  Week 12 (n=313,311,309,95) | 69.01 | 85.53 | 87.06 | 23.16

13. Secondary Outcome: Median Time to PASI50 Response During the 12-Week Double-Blind Treatment
Time Frame: Baseline up to Week 12
Population: FAS; OC
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 329 | 330 | 335 | 107
weeks | 8.1 [NA to NA] — The lower (upper) bound of the 95% confidence interval (CI) was not estimable because the lower (upper) bound of the survival function using LogLog transformation was not below the median. | 5.0 [4.1 to 8.0] | 7.9 [4.4 to 8.0] | NA [NA to NA] — Median and 95% CI were not estimable due to less than (<)50% of events occurring.

14. Secondary Outcome: Percentage of Participants Who Achieved a 90% Reduction in PASI Relative to Baseline (PASI90) During the 12-Week Double-Blind Treatment
Description: as for outcome 12
Time Frame: Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 326 | 327 | 331 | 106
percentage of participants
  Week 2 (n=326,327,331,106) | 0.00 | 0.61 | 0.30 | 0.00
  Week 4 (n=319,323,328,102) | 1.57 | 4.64 | 1.83 | 0.00
  Week 8 (n=315,319,323,99) | 12.06 | 26.02 | 15.79 | 0.00
  Week 12 (n=313,311,309,95) | 22.04 | 38.26 | 34.95 | 1.05

15. Secondary Outcome: Median Time to Achieve PASI75 Response During the 12-Week Double-Blind Treatment
Time Frame: Baseline up to Week 12
Population: FAS; OC
Measure: Median (95% Confidence Interval); unit: weeks
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 329 | 330 | 335 | 107
weeks | 12.6 [12.4 to 13.1] | 8.6 [8.1 to 12.1] | 12.1 [11.1 to 12.1] | NA [NA to NA] — Median and 95% CI were not estimable due to <50% of events occurring.

16. Secondary Outcome: Percentage of Participants With a PASI Score Greater Than or Equal to (≥)125% of the Baseline PASI Score During the 12-Week Double-Blind Treatment
Time Frame: Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 326 | 327 | 331 | 106
percentage of participants
  Week 2 (n=326,327,331,106) | 0.92 | 0.61 | 0.30 | 4.72
  Week 4 (n=319,323,328,102) | 2.19 | 0.93 | 0.91 | 8.82
  Week 8 (n=315,319,323,99) | 2.54 | 0.31 | 0.31 | 7.07
  Week 12 (n=313,311,309,95) | 2.88 | 0.32 | 0.97 | 7.37
  Overall (n=327,329,334,107) | 4.59 | 1.82 | 1.80 | 15.89

17. Secondary Outcome: Mean Itch Severity Item (ISI) Score During the 12-Week Double-Blind Treatment
Description: ISI assessed severity of itch (pruritus) due to psoriasis. ISI is a single item, horizontal numeric rating scale. Participants were asked to rate "your worst itching due to psoriasis over the past 24 hours" on a numeric rating scale anchored by the terms "No itching" (0) and "Worst possible itching" (10) at the ends.
Time Frame: Baseline, Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 305 | 308 | 305 | 107
score on a scale
  Baseline (n=305,308,305,107) | 5.19 (0.16) | 5.26 (0.16) | 5.23 (0.15) | 5.15 (0.27)
  Week 2 (n=325,322,330,105) | 3.47 (0.15) | 2.87 (0.14) | 3.90 (0.15) | 4.90 (0.30)
  Week 4 (n=318,323,328,101) | 2.92 (0.15) | 1.86 (0.13) | 2.97 (0.13) | 4.65 (0.31)
  Week 8 (n=313,315,320,100) | 2.11 (0.14) | 1.22 (0.11) | 2.06 (0.13) | 4.74 (0.32)
  Week 12 (n=312,309,311,95) | 1.98 (0.14) | 1.25 (0.12) | 1.72 (0.13) | 4.75 (0.32)

18. Secondary Outcome: Mean Change From Baseline in ISI Score During the 12-Week Double-Blind Treatment
Description: as for outcome 17
Time Frame: Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 303 | 300 | 301 | 105
score on a scale
  Week 2 | -1.73 (0.15) | -2.39 (0.14) | -1.22 (0.15) | -0.26 (0.22)
  Week 4 | -2.24 (0.18) | -3.43 (0.17) | -2.20 (0.15) | -0.44 (0.24)
  Week 8 | -3.01 (0.18) | -4.02 (0.17) | -3.13 (0.17) | -0.46 (0.26)
  Week 12 | -3.18 (0.18) | -3.96 (0.18) | -3.46 (0.19) | -0.43 (0.28)

19. Secondary Outcome: Percentage of Participants Achieving an ISI Score of 0 During the 12-Week Double-Blind Treatment
Description: as for outcome 17
Time Frame: Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 288 | 281 | 294 | 98
percentage of participants
  Week 2 | 10.42 | 13.88 | 10.54 | 1.02
  Week 4 | 15.66 | 34.28 | 14.09 | 2.13
  Week 8 | 29.45 | 47.83 | 28.67 | 6.38
  Week 12 | 31.64 | 51.85 | 40.07 | 6.74

20. Secondary Outcome: Mean Dermatology Life Quality Index (DLQI) Score During the 12-Week Double-Blind Treatment
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life.
Time Frame: Baseline and Weeks 4 and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 328 | 326 | 332 | 106
score on a scale
  Baseline (n=328,326,332,106) | 12.98 (0.39) | 13.32 (0.38) | 12.73 (0.38) | 12.27 (0.69)
  Week 4 (n=318,323,325,100) | 7.82 (0.36) | 5.95 (0.32) | 6.90 (0.35) | 10.51 (0.77)
  Week 12 (n=306,305,307,93) | 5.61 (0.36) | 3.47 (0.27) | 3.84 (0.30) | 10.33 (0.81)

21. Secondary Outcome: Mean Change From Baseline in DLQI Score During the 12-Week Double-Blind Treatment
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life. The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline.
Time Frame: Weeks 4 and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 317 | 319 | 322 | 99
score on a scale
  Week 4 (n=317,319,322,99) | -5.28 (0.35) | -7.43 (0.36) | -5.80 (0.33) | -1.64 (0.55)
  Week 12 (n=305,301,305,93) | -7.33 (0.43) | -9.72 (0.40) | -8.97 (0.40) | -1.85 (0.66)

22. Secondary Outcome: Mean DLQI Subscale Scores During the 12-Week Double-Blind Treatment
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much); higher scores indicate poor quality of life. The DLQI can be analyzed under 6 subscales by combining questions and is categorized as follows: symptoms and feelings (maximum score=6); daily activities (maximum score=6); leisure (maximum score=6); work and school (maximum score=3); personal relationships (maximum score=6); and treatment (maximum score=3).
Time Frame: Baseline and Weeks 4 and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 328 | 327 | 332 | 106
score on a scale
  Symptoms and Feelings,Baseline (n=328,327,332,106) | 3.44 (0.09) | 3.49 (0.08) | 3.47 (0.08) | 3.46 (0.16)
  Symptoms and Feelings, Week 4 (n=318,323,324,100) | 2.11 (0.08) | 1.63 (0.07) | 1.94 (0.07) | 2.92 (0.15)
  Symptoms and Feelings, Week 12 (n=306,304,307,93) | 1.60 (0.09) | 1.04 (0.07) | 1.16 (0.07) | 2.85 (0.17)
  Daily Activities,Baseline (n=327,327,332,106) | 2.76 (0.10) | 2.85 (0.09) | 2.76 (0.09) | 2.52 (0.16)
  Daily Activities, Week 4 (n=318,322,324,100) | 1.68 (0.08) | 1.30 (0.08) | 1.53 (0.08) | 2.28 (0.18)
  Daily Activities, Week 12 (n=306,305,306,93) | 1.19 (0.08) | 0.70 (0.07) | 0.79 (0.07) | 2.17 (0.19)
  Leisure, Baseline (n=326,326,330,106) | 2.52 (0.11) | 2.67 (0.11) | 2.57 (0.11) | 2.25 (0.17)
  Leisure, Week 4 (n=318,322,325,100) | 1.50 (0.09) | 1.14 (0.08) | 1.33 (0.09) | 1.84 (0.18)
  Leisure, Week 12 (n=306,305,307,93) | 1.09 (0.09) | 0.70 (0.07) | 0.71 (0.07) | 1.90 (0.19)
  Work and School,Baseline (n=328,327,331,106) | 1.12 (0.06) | 1.08 (0.06) | 1.06 (0.06) | 0.97 (0.11)
  Work and School, Week 4 (n=318,323,325,100) | 0.56 (0.05) | 0.46 (0.05) | 0.54 (0.05) | 0.81 (0.11)
  Work and School, Week 12 (n=306,304,307,92) | 0.41 (0.04) | 0.24 (0.04) | 0.32 (0.04) | 0.83 (0.12)
  Personal Relationships,Baseline(n=328,326,332,106) | 1.95 (0.11) | 1.98 (0.10) | 1.67 (0.10) | 1.89 (0.18)
  Personal Relationships, Week 4 (n=318,323,325,100) | 1.21 (0.09) | 0.90 (0.08) | 0.93 (0.08) | 1.64 (0.20)
  Personal Relationships, Week 12 (n=306,305,307,93) | 0.85 (0.09) | 0.48 (0.06) | 0.52 (0.07) | 1.65 (0.20)
  Treatment, Baseline(n=328,327,332,106) | 1.22 (0.06) | 1.24 (0.06) | 1.23 (0.06) | 1.18 (0.10)
  Treatment, Week 4 (n=318,323,325,100) | 0.76 (0.05) | 0.52 (0.04) | 0.65 (0.04) | 1.02 (0.11)
  Treatment, Week 12 (n=306,305,307,93) | 0.45 (0.04) | 0.31 (0.03) | 0.33 (0.04) | 0.95 (0.11)

23. Secondary Outcome: Mean Change From Baseline in DLQI Subscale Scores During the 12-Week Double-Blind Treatment
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much); higher scores indicate poor quality of life. The DLQI can be analyzed under 6 subscales by combining questions and is categorized as follows: symptoms and feelings (maximum score=6); daily activities (maximum score=6); leisure (maximum score=6); work and school (maximum score=3); personal relationships (maximum score=6); and treatment (maximum score=3). The minimally important difference for the DLQI has been estimated as a 2 to 5 point change from baseline.
Time Frame: Weeks 4 and 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 317 | 320 | 321 | 99
scores on a scale
  Symptoms and Feelings, Week 4 (n=317,320,321,99) | -1.34 (0.09) | -1.87 (0.08) | -1.53 (0.08) | -0.53 (0.15)
  Symptoms and Feelings, Week 12 (n=305,301,305,93) | -1.81 (0.10) | -2.41 (0.10) | -2.30 (0.10) | -0.62 (0.18)
  Daily Activities, Week 4 (n=316,319,321,99) | -1.13 (0.09) | -1.57 (0.09) | -1.21 (0.09) | -0.28 (0.15)
  Daily Activities, Week 12 (n=304,302,304,93) | -1.58 (0.10) | -2.14 (0.10) | -1.96 (0.10) | -0.34 (0.19)
  Leisure, Week 4 (n=316,318,320,99) | -1.03 (0.10) | -1.54 (0.10) | -1.24 (0.10) | -0.39 (0.15)
  Leisure, Week 12 (n=303,301,303,93) | -1.41 (0.11) | -1.95 (0.11) | -1.90 (0.11) | -0.31 (0.18)
  Work and School, Week 4 (n=317,320,321,99) | -0.56 (0.06) | -0.63 (0.06) | -0.52 (0.06) | -0.13 (0.10)
  Work and School, Week 12 (n=305,301,304,92) | -0.69 (0.07) | -0.86 (0.06) | -0.77 (0.07) | -0.12 (0.10)
  Personal Relationships, Week 4 (n=317,319,322,99) | -0.76 (0.09) | -1.09 (0.09) | -0.73 (0.08) | -0.18 (0.14)
  Personal Relationships, Week 12 (n=305,301,305,93) | -1.10 (0.11) | -1.46 (0.10) | -1.17 (0.09) | -0.20 (0.15)
  Treatment, Week 4 (n=317,320,322,99) | -0.47 (0.06) | -0.72 (0.06) | -0.58 (0.06) | -0.12 (0.10)
  Treatment, Week 12 (n=305,302,305,93) | -0.75 (0.06) | -0.91 (0.06) | -0.91 (0.06) | -0.24 (0.10)

24. Secondary Outcome: Percentage of Participants Achieving DLQI Response ≥5 During the 12-Week Double-Blind Treatment
Description: as for outcome 20
Time Frame: Weeks 4 and 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 279 | 283 | 282 | 82
percentage of participants
  Week 4 | 60.93 | 71.38 | 61.35 | 36.59
  Week 12 | 71.54 | 85.28 | 81.34 | 35.90

25. Secondary Outcome: Percentage of Participants Achieving DLQI Response ≤1 During the 12-Week Double-Blind Treatment
Description: as for outcome 20
Time Frame: Weeks 4 and 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 306 | 312 | 316 | 95
percentage of participants
  Week 4 | 13.07 | 21.79 | 15.51 | 7.37
  Week 12 | 33.22 | 51.36 | 47.18 | 8.89

26. Secondary Outcome: Median Time to DLQI Response
Description: The DLQI is a general dermatology questionnaire that consists of 10 items that assess health related quality of life (daily activities, personal relationships, symptoms and feelings, leisure, work and school, and treatment). The DLQI questions are rated by the participant as 0 (not at all/not relevant) to 3 (very much) with a total score range of 0 (best) to 30 (worst); higher scores indicate poor quality of life. DLQI Response was defined as a 5-point reduction in the total DLQI score.
Time Frame: Weeks 4 and 12
Population: Data were not analyzed as the endpoint of proportion of participants achieving a 5-point reduction from baseline in DLQI provided similar information.
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 0 | 0 | 0 | 0

27. Secondary Outcome: Mean Short Form 36 (SF-36) Mental Component Summary (MCS) and Physical Component Summary (PCS) Scores at Baseline and Week 12
Description: The SF-36 is a general health status questionnaire that assesses 8 domains of functional health and well being: Physical Functioning, Role Limitations due to Physical Health Problems, Bodily Pain, Social Functioning, Mental Health, Role Limitations due to Emotional Problems, Vitality, and General Health Perceptions. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). A PCS score and MCS score are based on a normalized sum of the 8 scale scores; PCS/MCS summary concept score = (raw score*10) plus 50. Higher scores indicate a better health related quality of life.
Time Frame: Baseline and Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 327 | 327 | 327 | 105
score on a scale
  Baseline Physical Health Score (n=327,327,327,105) | 47.4 (0.5) | 48.3 (0.5) | 47.5 (0.5) | 46.8 (1.0)
  Week 12 Physical Health Score (n=303,304,307,95) | 51.7 (0.5) | 53.6 (0.4) | 52.5 (0.5) | 47.8 (1.0)
  Baseline Mental Health Score (n=327,327,327,105) | 42.0 (0.6) | 41.2 (0.6) | 42.0 (0.7) | 39.8 (1.2)
  Week 12 Mental Health Score (n=303,304,307,95) | 47.0 (0.6) | 49.3 (0.5) | 47.8 (0.6) | 41.7 (1.3)

28. Secondary Outcome: Mean SF-36 Domain Scores at Baseline and Week 12
Description: The SF-36 is a general health status questionnaire that assesses 8 domains of functional health and well being: Physical Functioning, Role Limitations due to Physical Health Problems, Bodily Pain, Social Functioning, Mental Health, Role Limitations due to Emotional Problems, Vitality, and General Health Perceptions. The score for a section is an average of the individual question scores, which are scaled 0-100 (100=highest level of functioning). Higher scores indicate a better health related quality of life.
Time Frame: Baseline and Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 328 | 328 | 330 | 106
score on a scale
  Baseline Physical Functioning (n=328,328,330,106) | 48.3 (0.5) | 49.0 (0.5) | 48.6 (0.5) | 46.7 (1.1)
  Week 12 Physical Functioning (n=306,305,308,95) | 51.9 (0.5) | 53.1 (0.4) | 52.2 (0.4) | 48.1 (1.1)
  Baseline Role Physical (n=328,328,330,106) | 45.4 (0.6) | 45.9 (0.6) | 45.5 (0.6) | 44.4 (1.1)
  Week 12 Role Physical (n=307,305,308,95) | 50.5 (0.5) | 52.5 (0.4) | 51.2 (0.5) | 46.1 (1.1)
  Baseline Bodily Pain (n=328,329,331,107) | 44.5 (0.7) | 45.6 (0.7) | 44.0 (0.7) | 43.6 (1.2)
  Week 12 Bodily Pain (n=306,305,307,95) | 51.7 (0.6) | 54.6 (0.5) | 52.4 (0.6) | 45.7 (1.3)
  Baseline General Health (n=328,328,330,106) | 43.4 (0.5) | 42.8 (0.5) | 43.5 (0.6) | 42.4 (1.0)
  Week 12 General Health (n=305,304,308,95) | 46.2 (0.5) | 48.5 (0.5) | 47.9 (0.5) | 42.6 (1.0)
  Baseline Vitality (n=328,329,331,107) | 47.9 (0.5) | 48.5 (0.6) | 48.3 (0.5) | 46.5 (1.0)
  Week 12 Vitality (n=306,305,307,95) | 52.4 (0.5) | 54.4 (0.5) | 52.9 (0.5) | 47.9 (1.1)
  Baseline Social Functioning (n=328,329,331,107) | 41.6 (0.6) | 41.1 (0.6) | 42.3 (0.7) | 40.7 (1.2)
  Week 12 Social Functioning (n=306,305,307,95) | 47.8 (0.6) | 50.6 (0.5) | 49.3 (0.5) | 42.0 (1.2)
  Baseline Role-Emotional (n=328,329,331,107) | 43.2 (0.7) | 42.4 (0.7) | 43.1 (0.7) | 40.4 (1.3)
  Week 12 Role-Emotional (n=306,305,307,95) | 48.6 (0.5) | 50.2 (0.5) | 48.6 (0.6) | 43.3 (1.4)
  Baseline Mental Health (n=328,329,331,107) | 42.0 (0.6) | 41.5 (0.6) | 41.7 (0.7) | 39.5 (1.2)
  Week 12 Mental Health (n=306,305,307,95) | 46.6 (0.6) | 48.9 (0.5) | 47.5 (0.6) | 41.4 (1.2)
  Baseline Health Transition (n=328,329,331,107) | 3.2 (0.0) | 3.2 (0.0) | 3.1 (0.0) | 3.2 (0.1)
  Week 12 Health Transition (n=306,305,307,95) | 2.6 (0.0) | 2.6 (0.0) | 2.5 (0.0) | 3.0 (0.1)

29. Secondary Outcome: Mean Change From Baseline in SF-36 MCS and PCS Scores
Description: as for outcome 27
Time Frame: Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 301 | 302 | 301 | 93
score on a scale
  Physical Health Score | 4.1 (0.4) | 5.0 (0.5) | 5.2 (0.5) | 0.8 (0.7)
  Mental Health Score | 5.0 (0.6) | 7.6 (0.6) | 5.8 (0.6) | 1.5 (1.1)

30. Secondary Outcome: Mean Change From Baseline in SF-36 Domain Scores
Description: as for outcome 28
Time Frame: Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 305 | 304 | 304 | 94
score on a scale
  Physical Functioning | 3.5 (0.4) | 3.7 (0.4) | 3.7 (0.5) | 1.1 (0.8)
  Role Physical | 5.1 (0.5) | 6.3 (0.6) | 6.1 (0.5) | 1.3 (0.9)
  Bodily Pain | 7.0 (0.7) | 8.5 (0.6) | 8.6 (0.7) | 1.6 (1.0)
  General Health | 2.5 (0.5) | 5.5 (0.5) | 4.4 (0.5) | 0.2 (0.8)
  Vitality | 4.2 (0.5) | 5.4 (0.5) | 4.6 (0.5) | 1.3 (0.9)
  Social Functioning | 6.0 (0.7) | 9.2 (0.6) | 7.3 (0.6) | 0.7 (1.1)
  Role - Emotional | 5.4 (0.6) | 7.2 (0.6) | 5.8 (0.7) | 2.3 (1.2)
  Mental Health | 4.5 (0.6) | 7.0 (0.6) | 5.9 (0.6) | 1.4 (1.1)
  Health Transition | -0.5 (0.1) | -0.6 (0.1) | -0.6 (0.1) | -0.2 (0.1)

31. Secondary Outcome: Percentage of Participants in Each Patient Global Assessment of Psoriasis (PtGA) Category During the 12-Week Double-Blind Treatment
Description: The PtGA asks the participant to evaluate the overall cutaneous disease at that point in time on a single item, 5-point scale (0=clear; 1=almost clear; 2=mild; 3=moderate; 4=severe).
Time Frame: Baseline and Weeks 2, 4, and 8
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 328 | 328 | 330 | 107
percentage of participants
  Clear, Baseline (n=328,328,330,107) | 0.0 | 0.0 | 0.0 | 0.0
  Almost Clear, Baseline (n=328,328,330,107) | 0.0 | 0.3 | 0.3 | 0.0
  Mild, Baseline (n=328,328,330,107) | 3.4 | 1.5 | 4.2 | 3.7
  Moderate, Baseline (n=328,328,330,107) | 32.3 | 30.2 | 28.5 | 23.4
  Severe, Baseline (n=328,328,330,107) | 64.3 | 68.0 | 67.0 | 72.9
  Clear, Week 2 (n=324,322,331,106) | 0.3 | 0.0 | 0.3 | 0.0
  Almost Clear, Week 2 (n=324,322,331,106) | 1.2 | 4.3 | 1.2 | 0.9
  Mild, Week 2 (n=324,322,331,106) | 13.3 | 14.9 | 11.8 | 2.8
  Moderate, Week 2 (n=324,322,331,106) | 49.4 | 54.3 | 52.0 | 38.7
  Severe, Week 2 (n=324,322,331,106) | 35.8 | 26.4 | 34.7 | 57.5
  Clear, Week 4 (n=319,323,324,100) | 0.3 | 0.6 | 0.3 | 0.0
  Almost Clear, Week 4 (n=319,323,324,100) | 6.9 | 17.0 | 9.3 | 0.0
  Mild, Week 4 (n=319,323,324,100) | 21.6 | 30.7 | 26.5 | 5.0
  Moderate, Week 4 (n=319,323,324,100) | 46.7 | 36.8 | 43.5 | 35.0
  Severe, Week 4 (n=319,323,324,100) | 24.5 | 14.9 | 20.4 | 60.0
  Clear, Week 8 (n=313,317,315,97) | 2.9 | 4.7 | 3.5 | 0.0
  Almost Clear, Week 8 (n=313,317,315,97) | 16.9 | 38.2 | 29.8 | 4.1
  Mild, Week 8 (n=313,317,315,97) | 33.5 | 27.1 | 33.0 | 7.2
  Moderate, Week 8 (n=313,317,315,97) | 31.3 | 22.1 | 24.8 | 38.1
  Severe, Week 8 (n=313,317,315,97) | 15.3 | 7.9 | 8.9 | 50.5

32. Secondary Outcome: Percentage of Participants With a PtGA Response During the 12-Week Double-Blind Treatment
Description: The PtGA asks the participant to evaluate the overall cutaneous disease at that point in time on a single item, 5-point scale (0=clear; 1=almost clear; 2=mild; 3=moderate; 4=severe). Response defined as score of 0 or 1.
Time Frame: Weeks 2, 4, 8, and 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 324 | 322 | 331 | 106
percentage of participants
  Week 2 (n=324,322,331,106) | 1.54 | 4.35 | 1.51 | 0.94
  Week 4 (n=319,323,324,100) | 7.21 | 17.65 | 9.57 | 0.00
  Week 8 (n=313,317,315,97) | 19.81 | 42.90 | 33.33 | 4.12
  Week 12 (n=306,304,309,95) | 32.68 | 56.25 | 53.07 | 1.05

33. Secondary Outcome: Percentage of Participants in Each Patient Satisfaction With Study Medication (PSSM) Category During the 12-Week Double-Blind Treatment
Description: The PSSM is a single, 7 point item that evaluates overall participant satisfaction with the study treatment. Response options range from "very dissatisfied" to "very satisfied" with the study medication.
Time Frame: Week 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 307 | 305 | 306 | 95
percentage of participants
  Very satisfied | 44.0 | 68.5 | 62.4 | 15.8
  Somewhat satisfied | 27.0 | 17.4 | 23.5 | 15.8
  Slightly satisfied | 11.7 | 5.2 | 7.2 | 11.6
  Neither satisfied nor dissatisfied | 4.6 | 2.3 | 2.0 | 11.6
  Slightly dissatisfied | 2.6 | 1.6 | 2.0 | 4.2
  Somewhat dissatisfied | 4.6 | 3.0 | 2.0 | 12.6
  Very dissatisfied | 5.5 | 2.0 | 1.0 | 28.4

34. Secondary Outcome: Percentage of Participants Achieving PSSM Response of 'Very Satisfied' or 'Somewhat Satisfied' at Week 12
Description: as for outcome 33
Time Frame: Week 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 307 | 305 | 306 | 95
percentage of participants | 71.01 | 85.90 | 85.95 | 31.58

35. Secondary Outcome: Mean European Quality of Life 5 Dimension (EQ-5D) Health State Utility Score During the 12-Week Double-Blind Treatment
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 domains: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed"). Scoring formula developed by EuroQol Group assigns a utility value for each domain in the profile. Score is transformed and results in a total score range -0.594 to 1.000; higher score indicates a better health state.
Time Frame: Baseline and Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 325 | 326 | 330 | 104
score on a scale
  Baseline | 0.7 (0.0) | 0.7 (0.0) | 0.7 (0.0) | 0.6 (0.0)
  Week 12 | 0.8 (0.0) | 0.9 (0.0) | 0.9 (0.0) | 0.7 (0.0)

36. Secondary Outcome: Least Squares (LS) Mean Change From Baseline in EQ-5D Health State Utility Score During the 12-Week Double-Blind Treatment
Description: as for outcome 35
Time Frame: Week 12
Population: FAS; OC
Measure: Least Squares Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 301 | 300 | 303 | 92
scores on a scale | 0.14 (0.011) | 0.21 (0.011) | 0.19 (0.011) | 0.03 (0.021)

37. Secondary Outcome: Mean EQ-5D Visual Analog Score (VAS) During the 12-Week Double-Blind Treatment
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single index value. The VAS component rates current health state on a scale from 0 mm (worst imaginable health state) to 100 mm (best imaginable health state); higher scores indicate a better health state.
Time Frame: Baseline and Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: mm
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 315 | 318 | 312 | 100
mm
  Baseline (n=315,318,312,100) | 63.3 (1.3) | 63.3 (1.3) | 64.2 (1.3) | 60.5 (2.7)
  Week 12 (n=298,294,297,91) | 75.3 (1.1) | 81.1 (1.0) | 80.0 (1.0) | 65.1 (2.6)

38. Secondary Outcome: Mean Change From Baseline in EQ-5D VAS at Week 12
Description: as for outcome 37
Time Frame: Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: mm
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 289 | 288 | 285 | 88
mm | 11.6 (1.4) | 16.6 (1.5) | 15.7 (1.4) | 3.0 (2.4)

39. Secondary Outcome: Dimension Health State EQ-5D Score During the 12-Week Double-Blind Treatment
Description: EQ-5D: participant rated questionnaire to assess health-related quality of life in terms of a single utility score. Health State Profile component assesses level of current health for 5 dimensions: mobility, self-care, usual activities, pain and discomfort, and anxiety and depression. The score for each of the 5 dimensions can range from 1 to 3; 1 indicates better health state (no problems); 3 indicates worst health state ("confined to bed").
Time Frame: Baseline and Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: Units on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 326 | 327 | 330 | 104
Units on a scale
  Mobility, Baseline (n=326,327,330,104) | 1.3 (0.0) | 1.3 (0.0) | 1.3 (0.0) | 1.3 (0.0)
  Mobility, Week 12 (n=306,304,307,95) | 1.2 (0.0) | 1.1 (0.0) | 1.2 (0.0) | 1.3 (0.1)
  Self Care, Baseline (n=327,327,330,104) | 1.2 (0.0) | 1.1 (0.0) | 1.1 (0.0) | 1.2 (0.0)
  Self Care, Week 12 (n=306,304,307,95) | 1.1 (0.0) | 1.0 (0.0) | 1.1 (0.0) | 1.2 (0.0)
  Usual Activities, Baseline (n=327,327,330,104) | 1.4 (0.0) | 1.4 (0.0) | 1.4 (0.0) | 1.5 (0.1)
  Usual Activities, Week 12 (n=307,304,307,95) | 1.2 (0.0) | 1.1 (0.0) | 1.2 (0.0) | 1.3 (0.1)
  Pain/Discomfort, Baseline (n=327,328,330,104) | 1.8 (0.0) | 1.8 (0.0) | 1.9 (0.0) | 1.8 (0.1)
  Pain/Discomfort, Week 12 (n=307,304,307,95) | 1.5 (0.0) | 1.3 (0.0) | 1.4 (0.0) | 1.7 (0.1)
  Anxiety/Depression, Baseline (n=326,327,330,104) | 1.6 (0.0) | 1.7 (0.0) | 1.6 (0.0) | 1.7 (0.1)
  Anxiety/Depression, Week 12 (n=305,304,307,95) | 1.4 (0.0) | 1.3 (0.0) | 1.3 (0.0) | 1.5 (0.1)

40. Secondary Outcome: Mean Change From Baseline in EQ-5D Dimension Health State Score at Week 12
Description: as for outcome 39
Time Frame: Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 305 | 302 | 303 | 92
scores on a scale
  Mobility | -0.1 (0.0) | -0.1 (0.0) | -0.1 (0.0) | -0.0 (0.0)
  Self-Care | -0.1 (0.0) | -0.1 (0.0) | -0.1 (0.0) | -0.1 (0.0)
  Usual Activities | -0.3 (0.0) | -0.3 (0.0) | -0.2 (0.0) | -0.1 (0.1)
  Pain/Discomfort | -0.4 (0.0) | -0.5 (0.0) | -0.5 (0.0) | -0.1 (0.1)
  Anxiety/Depression | -0.2 (0.0) | -0.4 (0.0) | -0.3 (0.0) | -0.1 (0.1)

41. Secondary Outcome: Percentage of Participants Interacting With Healthcare Professionals During the 12-Week Double-Blind Treatment
Description: The Psoriasis Health Care Resource Utilization (Ps-HCRU) questionnaire is a short questionnaire designed to assess healthcare resource use and the impact of psoriasis on work. The first section assesses direct costs associated with healthcare resource use (interactions with healthcare providers such as general practitioners [GPs], primary care physicians [PCPs], or family medicine physicians [FMP], emergency room visits, and hospitalizations), and the second section assesses indirect costs associated with absenteeism due to psoriasis and the impact of psoriasis on productivity at work.
Time Frame: Baseline (BL) and Week 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 255 | 251 | 261 | 79
percentage of participants
  Baseline, GP/PCP/FMP (n=230,220,224,77) | 0.8 | 0.9 | 1.3 | 2.5
  Baseline, Dermatologist (n=230,220,224,77) | 6.9 | 4.5 | 7.5 | 10.3
  Baseline, Rheumatologist (n=230,220,224,77) | 0.0 | 0.0 | 0.0 | 0.0
  Baseline, Cardiologist (n=230,220,224,77) | 0.4 | 0.4 | 0.4 | 2.5
  Baseline, Gastroenterologist (n=230,220,224,77) | 0.4 | 0.0 | 0.0 | 0.0
  Baseline, Psychiatrist (n=230,220,224,77) | 0.0 | 0.4 | 0.0 | 1.2
  Baseline, Surgeon (n=230,220,224,77) | 0.4 | 0.0 | 0.0 | 0.0
  Baseline, Nurse (n=230,220,224,77) | 1.3 | 1.3 | 0.8 | 2.5
  Baseline, Other (n=230,220,224,77) | 2.1 | 0.9 | 0.0 | 1.2
  Week 12, GP/PCP/FMP (n=255,251,261,79) | 10.1 | 6.7 | 8.4 | 8.8
  Week 12, Dermatologist (n=255,251,261,79) | 8.2 | 4.3 | 5.7 | 7.5
  Week 12, Rheumatologist (n=255,251,261,79) | 0.7 | 1.1 | 0.7 | 0.0
  Week 12, Cardiologist (n=255,251,261,79) | 1.5 | 1.9 | 2.6 | 1.2
  Week 12, Gastroenterologist (n=255,251,261,79) | 1.1 | 1.5 | 1.5 | 0.0
  Week 12, Psychiatrist (n=255,251,261,79) | 0.0 | 0.7 | 1.5 | 0.0
  Week 12, Surgeon (n=255,251,261,79) | 0.3 | 0.3 | 0.0 | 0.0
  Week 12, Nurse (n=255,251,261,79) | 1.1 | 1.9 | 2.6 | 0.0
  Week 12, Other (n=255,251,261,79) | 8.6 | 5.1 | 6.8 | 2.5

42. Secondary Outcome: Percentage of Participants Reporting Healthcare Resource Use Events During the 12-Week Double-Blind Treatment
Time Frame: Week 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 230 | 225 | 238 | 71
percentage of participants | 10.43 | 9.78 | 10.08 | 8.45

43. Secondary Outcome: Percentage of Participants Employed or Not Employed and the Impact of Psoriasis on Work
Description: Psoriasis Health Care Resource Utilization Questionnaire is a short questionnaire designed to assess healthcare resource use and the impact of psoriasis on work. The questionnaire assesses employment status of participant (employed: yes or no) and if currently employed it asks the participant if they were absent or on sick leave from work due to psoriasis; if unemployed it asks the participant if the unemployment is due to psoriasis.
Time Frame: Baseline and Week 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 230 | 219 | 224 | 77
percentage of participants
  Baseline, employed | 67.8 | 71.2 | 72.3 | 71.4
  Baseline, absent/sick leave due to psoriasis | 18.3 | 21.0 | 22.3 | 23.4
  Baseline, not employed | 32.2 | 28.8 | 27.7 | 28.6
  Baseline, unemployed due to psoriasis | 9.6 | 7.3 | 6.3 | 2.6
  Week 12, employed | 69.2 | 73.8 | 69.1 | 68.1
  Week 12, absent/sick leave due to psoriasis | 13.2 | 14.7 | 15.7 | 17.4
  Week 12, not employed | 30.8 | 26.2 | 30.9 | 31.9
  Week 12, unemployed due to psoriasis | 4.0 | 4.9 | 4.7 | 4.3

44. Secondary Outcome: Percentage of Participants Reporting Work-Impacted Events During the 12-Week Double-Blind Treatment
Description: Psoriasis Health Care Resource Utilization Questionnaire is a short questionnaire designed to assess healthcare resource use and the impact of psoriasis on work.
Time Frame: Week 12
Population: FAS; OC
Measure: Number; unit: percentage of participants
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 158 | 164 | 164 | 48
percentage of participants | 37.97 | 30.49 | 34.15 | 56.25

45. Secondary Outcome: Mean Psoriasis Quality of Life 12 (PQOL-12) Score During the 12-Week Double-Blind Treatment
Description: The PQOL-12 is a 12-item questionnaire; 8 of the items on the Koo-Menter Psoriasis Index 12-item Quality of Life Questionnaire (PQOL-12) focus on emotional issues associated with psoriasis (self conscious, helpless, embarrassed, ability to enjoy life). The last 4 items deal with physical symptoms (pain or soreness, itch, physical irritation) and choice of clothing. The recall period is over the past month. The questions are answered on a scale from 0 to 10 with 0 being best and 10 being worst. Scores from each question are summed to give a total score (range 0 -120); higher scores indicate greater impairment to quality of life.
Time Frame: Baseline and Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 323 | 326 | 331 | 105
score on a scale
  Baseline (n=323,326,331,105) | 75.4 (1.5) | 77.0 (1.5) | 75.7 (1.5) | 74.9 (2.9)
  Week 12 (n=303,303,306,92) | 40.0 (1.8) | 29.2 (1.6) | 31.0 (1.7) | 65.5 (3.5)

46. Secondary Outcome: Mean Change From Baseline in PQOL-12 Score During the 12-Week Double-Blind Treatment
Description: The PQOL-12 is a 12-item questionnaire; 8 of the items on the PQOL-12) focus on emotional issues associated with psoriasis (self conscious, helpless, embarrassed, ability to enjoy life). The last 4 items deal with physical symptoms (pain or soreness, itch, physical irritation) and choice of clothing. The recall period is over the past month. The questions are answered on a scale from 0 to 10 with 0 being best and 10 being worst. Scores from each question are summed to give a total score (range 0 -120); higher scores indicate greater impairment to quality of life.
Time Frame: Week 12
Population: FAS; OC
Measure: Mean (Standard Error); unit: scores on a scale
Arm/Group | CP-690,550 5 mg Twice Daily (BID)+Placebo Twice Weekly (BIW) | CP-690,550 10 mg BID + Placebo BIW | Placebo BID + Etanercept 50 mg BIW | Placebo BID + Placebo BIW
Number analyzed (Participants) | 299 | 299 | 303 | 90
scores on a scale | -35.2 (1.9) | -47.9 (1.8) | -44.3 (1.8) | -9.6 (2.6)

ADVERSE EVENTS:
Description: The same event may appear as both an adverse event (AE) and a serious adverse event (SAE). However, what is presented are distinct events. An event may be categorized as serious in one subject and as nonserious in another subject, or one subject may have experienced both a serious and nonserious event during the study.
Groups:
- CP-690,550 5 mg BID: Participants received CP-690,550 5 mg tablets, orally, BID at approximately 12-hour intervals and placebo SC injections BIW at approximately 3- to 4-day intervals for 12 weeks.
- CP-690,550 10 mg BID: Participants received CP-690,550 10 mg tablets, orally, BID at approximately 12-hour intervals and placebo SC injections BIW at approximately 3- to 4-day intervals for 12 weeks.
- Etanercept 50 mg BIW: Participants received matching placebo tablets, orally, BID at approximately 12-hour intervals and etanercept 50 mg SC injections BIW at approximately 3- to 4-day intervals for 12 weeks.
- Placebo: Participants received matching placebo tablets, orally, BID at approximately 12-hour intervals and placebo SC injections BIW at approximately 3- to 4-day intervals for 12 weeks.
Arm/Group | CP-690,550 5 mg BID | CP-690,550 10 mg BID | Etanercept 50 mg BIW | Placebo
Serious Adverse Events (participants affected / at risk) | 7/329 | 5/330 | 7/335 | 2/107
Other Adverse Events (participants affected / at risk) | 103/329 | 121/330 | 109/335 | 34/107
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg BID (N=329) | CP-690,550 10 mg BID (N=330) | Etanercept 50 mg BIW (N=335) | Placebo (N=107)
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0 | 0
Uveitis (Eye disorders) | 0 | 0 | 1 | 0
Oedema peripheral (General disorders) | 0 | 0 | 0 | 1
Jaundice (Hepatobiliary disorders) | 0 | 0 | 1 | 0
Bronchitis (Infections and infestations) | 0 | 0 | 1 | 0
Diverticulitis (Infections and infestations) | 1 | 0 | 0 | 0
Extradural abscess (Infections and infestations) | 1 | 0 | 0 | 0
Paronychia (Infections and infestations) | 0 | 1 | 0 | 0
Perineal abscess (Infections and infestations) | 0 | 0 | 1 | 0
Pneumonia (Infections and infestations) | 0 | 1 | 0 | 0
Foot fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lower limb fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Poisoning (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Ischaemic cerebral infarction (Nervous system disorders) | 0 | 0 | 1 | 0
Depression (Psychiatric disorders) | 1 | 0 | 0 | 0
Renal colic (Renal and urinary disorders) | 1 | 0 | 0 | 0
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Psoriasis (Skin and subcutaneous tissue disorders) | 0 | 2 | 1 | 2
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | CP-690,550 5 mg BID (N=329) | CP-690,550 10 mg BID (N=330) | Etanercept 50 mg BIW (N=335) | Placebo (N=107)
Abdominal pain upper (Gastrointestinal disorders) | 3 | 1 | 7 | 2
Diarrhoea (Gastrointestinal disorders) | 8 | 7 | 7 | 3
Injection site erythema (General disorders) | 0 | 1 | 18 | 0
Injection site reaction (General disorders) | 0 | 0 | 12 | 0
Folliculitis (Infections and infestations) | 1 | 2 | 3 | 3
Nasopharyngitis (Infections and infestations) | 21 | 30 | 25 | 10
Upper respiratory tract infection (Infections and infestations) | 6 | 4 | 7 | 0
Urinary tract infection (Infections and infestations) | 4 | 3 | 5 | 3
Blood cholesterol increased (Investigations) | 9 | 11 | 7 | 0
Blood creatine phosphokinase increased (Investigations) | 15 | 16 | 10 | 0
Dyslipidaemia (Metabolism and nutrition disorders) | 10 | 15 | 3 | 1
Hypercholesterolaemia (Metabolism and nutrition disorders) | 11 | 14 | 5 | 2
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 10 | 4 | 1
Headache (Nervous system disorders) | 21 | 24 | 13 | 4
Cough (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 1 | 3
Psoriasis (Skin and subcutaneous tissue disorders) | 3 | 1 | 2 | 4
Hypertension (Vascular disorders) | 7 | 6 | 6 | 0

LIMITATIONS AND CAVEATS:
Clinical interpretation regarding sub-phenotypes of psoriasis (e.g., scalp psoriasis) should not be made based on the reported assessments by body regions. For example, the body region of head does not reflect solely scalp psoriasis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.